CLINICAL TRIAL: NCT02038348
Title: Interest of the 18F-DOPA-PET Imaging in Metastatic Melanoma Treated With B-RAF Inhibitors: a Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013-003294-10; 2013-35 (Other: AP HM)
Record Dates: First submitted 2013-12-03; First posted 2014-01-16 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET with 18F-FDOPA (Other)
  Interventions: Device: PET with 18F-FDOPA

INTERVENTIONS:
Device: PET with 18F-FDOPA

SUMMARY:
Melanoma incidence is increasing in most developed countries. At the metastatic stage, the prognosis is usually poor. Major advances have been obtained over the last 3 years with the development of therapies targeting the MAP kinases pathway.

Vemurafenib (zelboraf®) is approved in France since 2012 as first treatment of metastatic melanoma carrying a B-RAF mutation.

For growth, the tumor needs an adequate supply of nutrients to allow the synthesis of macromolecules and a contribution in carbon elements to ensure the production of energy. The nutrition demand is met through greater availability of nutrients via tumor angiogenesis and through increased intracellular penetration of nutrients via specific upregulation of transport systems and metabolic pathways.

Scanner is the imaging method most commonly used for the evaluation of therapeutic response. Such a method gives a morphological indication but does not evaluate the metabolic response.

With the development of functional imaging techniques and the advent of positron emission tomography (PET), it is now possible to obtain an assessment of the metabolic activity of tumors. The use of 18F-FDG to assess therapeutic responses to targeted therapies is fairly recent. The advantage of this approach is well documented for GIST and non-small cell lung cancer. In melanoma, the metabolic response to 18F-FDG is much faster than the response to TAP scanner.

18F-FDG tracer that targets glucose metabolism, is the most sensitive functional imaging in melanoma, which has hindered the development of other tracers such as 18F-FDOPA and 18F-FLT. The 18F-FDG TEP can thus be used in the initial staging and follow-up of the disease, a situation in which it can replace the TAP scanner, additional brain imaging remaining necessary.

The use of metabolic imaging to study the response to targeted therapies in melanoma has been the subject of only one publications. There was a trend toward improved progression-free survival in patients with high metabolic response at day J15.

For melanoma, the diagnostic sensitivity of PET 18F-FDOPA is lower than that of 18F-FDG (64% versus 95%). In contrast, the 18F-FDOPA tracer has the advantage of allowing a brain assessment, which is critical in melanoma that gives frequent metastases in the central nervous system. There has never been any evaluation of the metabolic response to targeted therapies such as BRAF inhibitors PET with 18F-FDOPA.

The investigators propose to conduct a monocentric prospective preliminary study to explore the potential usefulness of the metabolic PET imaging with 18F-FDOPA in the evaluation of metabolic response of B-RAF mutated metastatic melanoma treated with vemurafenib.

ELIGIBILITY:
Inclusion Criteria:

* B-RAF mutated metastatic melanoma.
* Reference imaging <1 month inclduing a whole body CT and 18F-FDG.
* At least one metastatic lesion at least with a diameter> 10 mm on CT.
* To which the staff has proposed, a B-RAF inhibitor in first-line treatment
* Signed informed consent.

Exclusion Criteria:

* Minor subject.
* Subject diabetic.
* Women of childbearing potential without effective contraception, with positive pregnancy test.
* Other known active cancer.
* No affiliation to a social security (beneficiary or assignee).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2016-02-16 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
brain metastases metabolic profile obtained with PET 18F-FDOPA | 24 MONTHS
  The profiles of metabolic changes in volume (expressed in%) obtained with each of the two tracers in conjunction with morphological volume changes observed on CT scan for non-brain metastases and brain metastases, respectively, will determine in first approach

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France